CLINICAL TRIAL: NCT04531982
Title: A Phase 3, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Pimavanserin as Adjunctive Treatment for the Negative Symptoms of Schizophrenia
Brief Title: Efficacy and Safety of Pimavanserin as Adjunctive Treatment for the Negative Symptoms of Schizophrenia
Acronym: ADVANCE-2
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: ACADIA Pharmaceuticals Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACP-103-064
Record Dates: First submitted 2020-08-26; First posted 2020-08-31 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — pimavanserin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Drug - Pimavanserin (Experimental): Pimavanserin 34 mg taken as two tablets + background antipsychotic, once daily by mouth
  Interventions: Drug: Pimavanserin
- Placebo (Placebo Comparator): Placebo + background antipsychotic, taken as two tablets, once daily by mouth
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pimavanserin — Pimavanserin 34 mg, taken as two blinded 17 mg tablets once daily by mouth
  Arms: Drug - Pimavanserin
Drug: Placebo — Placebo, taken as two blinded tablets once daily by mouth
  Arms: Placebo

SUMMARY:
To evaluate the efficacy and safety of adjunctive pimavanserin compared with adjunctive placebo in the treatment of negative symptoms of schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ≥18 and ≤55 years of age at the time of Screening
* Has a caregiver or some other identified responsible person (e.g., family member, social worker, caseworker, or nurse) considered reliable by the Investigator in providing support to the subject to help ensure compliance with study treatment, study visits, and protocol procedures, and who is also able to provide input helpful for completing study rating scales
* Diagnosis of schizophrenia made ≥1 year prior to Screening
* Is being treated must be one of the antipsychotics listed below:

  * Aripiprazole

    * Aripiprazole long-acting injectables
    * Abilify Maintena®
  * Aristada®
  * Asenapine
  * Brexpiprazole
  * Cariprazine
  * Lurasidone
  * Olanzapine
  * Paliperidone extended release (ER) (≤9 mg)
  * Paliperidone palmitate

    * Invega Sustenna® (≤156 mg)
    * Invega Trinza® (≤546 mg)
    * Trevicta® (≤350 mg)
    * Xeplion® (≤100 mg)
  * Risperidone
  * Risperidone long-acting injection
* Must be medically stable (including no recent hospitalization for exacerbation of psychiatric disorder) and has been medically stable for at least 12 weeks prior to Screening, in the opinion of the Investigator

Exclusion Criteria:

* Has a current comorbid psychiatric disorder other than schizophrenia or a disorder that would interfere with the ability to complete study assessments
* Is at a significant risk of suicide, in the opinion of the Investigator
* Has a significant risk of violent behavior in the opinion of the Investigator
* A confirmed urine drug screen (UDS) result at Baseline that indicates the presence of any tested prohibited substance of potential abuse, including marijuana
* Is taking a medication or drug or other substance that is prohibited according to this protocol, including medications that prolong the QT interval, strong cytochrome P450 (CYP) 3A4 enzyme (CYP3A4) inhibitors and inducers
* Known family or personal history or symptoms of long QT syndrome or risk factors for torsade de pointes and/or sudden death, including symptomatic bradycardia, hypokalemia or hypomagnesemia, and the presence of congenital prolongation of the QT interval
* Current evidence, or history within the previous 12 weeks prior to Screening, of a serious and/or unstable psychiatric, neurologic, cardiovascular, respiratory, gastrointestinal, renal, hepatic, hematologic, or other medical disorder, including cancer or malignancies that in the judgment of the Investigator would jeopardize the safe participation of the subject in the study
* Has moderate to severe congestive heart failure
* Has a history of myocardial infarction within 6 months prior to enrollment
* Has a body mass index (BMI) <19 or ≥35 at Screening

Additional inclusion/exclusion criteria apply. Patients will be evaluated at screening to ensure that all criteria for study participation are met. Patients may be excluded from the study based on these assessments (and specifically, if it is determined that their baseline health and condition do not meet all prespecified entry criteria).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 454 (Actual)
Dates: Start 2020-08-05 (Actual); Primary Completion 2024-01-25 (Actual); Study Completion 2024-02-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (102):
- Argentina (11):
  - 603-Fundación para el Estudio y Tratamiento de las Enfermedades Mentales - FETEM, Buenos Aires
  - 610-Clinica Privada Banfield S.A., Buenos Aires
  - 625-NOVAIN Neurociencias Group, Buenos Aires
  - 601-CENydET- Centro Neurobiologico y de Estres Traumatico-Biopsychomedical Research Group SRL, Ciudad Autonoma Buenos Aires
  - 602-FunDamoS, Ciudad Autonoma Buenos Aires
  - 622-Instituto Medico Damic Srl, Córdoba
  - 624-Centro Especializado en Neurociencias CEN, Córdoba
  - 626-Sanatorio Prof. Leon S. Morra S.A., Córdoba
  - 617-INSA Instituto de Neurociencias San Agustin S.A., La Plata
  - 623-Clinica Privada de Salud Mental Santa Teresa de Avila, La Plata
  - 607-Resolution Psicopharmacology Research Institute, Mendoza
- Bulgaria (17):
  - 532-MHAT "Dr. Hristo Stambolski", EOOD, Kazanlak, Stara Zagora
  - 454-Mental Health Center Prof. Dr. Ivan Temkov - Burgas EO Burgas; Department for Treatment of Emergency Psychiatric Conditions, Burgas
  - 533-State Psychiatric Hospital - Kardzhali, EOOD, Kardzhali
  - 569-State Psychiatric Hospital - Lovech, Lovech
  - 535-UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - 586-Medical Center Mentalcare OOD, Plovdiv
  - 563-MC-Hipokrat-N E00D, Plovdiv
  - 592-Medical center Spectar - Plovdiv EOOD, Plovdiv
  - 570-Medical Centre "Sveti Naum", Sofia
  - 526-DCC "Sv. Vrach and Sv. Sv. Kuzma and Damyan", OOD, Sofia
  - 405-"UMHAT Alexandrovska EAD, Sofia; Clinic of Psychiatry, First Department of Psychiatry ", Sofia
  - 568-Medical Center Hera EOOD, Sofia
  - 528-Medical Center Intermedica, OOD, Sofia
  - 590-State Psychiatric Hospital - Tzarev Brod, Tsarev Brod
  - 498-DCC "Mladost M" - Varna, OOD, Varna
  - 455-Mental Health Center - Veliko Tarnovo EOOD,, Veliko Tarnovo
  - 401-Mental Health Center - Vratsa EOOD, Vratsa; Department of Psychiatry, Vratsa
- Croatia (5):
  - 536-Clinic for psychiatry Vrapce, Zagreb
  - 537-Clinic for psychiatry Vrapce, Zagreb
  - 550-Clinic for psychiatry Vrapce, Zagreb
  - 557-Clinic for psychiatry Vrapce, Zagreb
  - 594-klinika za psihijatriju Sveti Ivan, n/p Igor Filipčić or Marija Zelenika, Zagreb
- Czechia (5):
  - 512-NeuropsychiatrieHK s.r.o., Hradec Králové
  - 583-Narodni ustav dusevniho zdravi, Klecany
  - 519-A-SHINE s.r.o., Pilsen
  - 513-CLINTRIAL s.r.o., Prague
  - 499-MUDr. Tibor Miklos, Prague
- Hungary (4):
  - 410-Mathe es Tarsa Bt., Kalocsa, Bacs
  - 456-Semmelweis University Department of Psychiatry and Psychotherapy, Budapest
  - 520-Nyiro Gyula Korhaz - Orszagos Pszichiatriai es Addiktologiai Intezet, Budapest
  - 440-PsychoTech Kft., Pécs
- Italy (4):
  - 580-AOU Consorziale Policlinico di Bari, Bari
  - 539-"Fondazione IRCCS CA' Granda Ospedale Maggiore Policlinico U.O.C. Psichiatria - Padiglione Alfieri, primo piano", Milan
  - 566-Ospedale San Raffaele (San Raffaele Turro), Milan
  - 553-AO Città della Salute e della Scienza di Torino, Torino
- Lithuania (4):
  - 516-Neuromeda, JSC, Kaunas
  - 483-Romuvos klinika, UAB, Kaunas
  - 518-Kaunas City Outpatient Clinic, Public Institution, Kaunas
  - 484-Medical Center Puriena JSC, Šilutė
- Poland (7):
  - 525-Podlaskie Centrum Psychogeriatrii, Bialystok
  - 502-Przychodnia Srodmiescie Sp. z o. o., Bydgoszcz
  - 579-Centrum Badan Klinicznych P.I. House Sp. z o.o., Gdansk
  - 541-Care Clinic centrum Medyczne, Katowice
  - 501-Specjalistyczna Praktyka Lekarska Marek Domański, Lublin
  - 578-MSCZ im. prof. J. Mazurkiewicza, Pruszków
  - 540-Ośr. Badań Klin. CLINSANTE S.C., Torun
- Russia (18):
  - 417-State budget healthcare Institution of Stavropol region "Regional specialized psychiatric hospital #2"., Tonnel’nyy, Stavropol Kray
  - 505-GUZ Lipetsk Regional psychoneurological Hospital #1, Lipetsk
  - 573-"SBIH of Moscow ""Psychiatric Clinical Hospital # 4 n.a. P.B. Gannushkin"" Short name: PCH N4 n.a. P.B.Gannushkin", Moscow
  - 581-SBIH of Moscow "Psych Clinical Hospital #1 N.A. Alekseev", Moscow
  - 415-Saint-Petersburg state healthcare institution "Saint Nicolas wonderworker psychiatric hospital", Saint Petersburg
  - 571-St. Petersburg SHI "Psychoneurological Dispensary #10", Saint Petersburg
  - 451-V. M. Bekhterev National Research Medical Center For Psychiatry and Neurology, Saint Petersburg
  - 453-"Saint-Petersburg Scientific Research Psychoneurological Institute n.a. V.M. Bekhterev", Saint Petersburg
  - 465-"Saint-Petersburg Scientific Research Psychoneurological Institute n.a. V.M. Bekhterev, Saint Petersburg
  - 495-"FSBI "National medical scientific center of psychiatry and neurology n.a. V.M. Bekhterev" MoH Short name: NMSC of Psy&Neuro n.a. Bekhterev, 12 dep.", Saint Petersburg
  - 464-Saint Petersburg State Budget Healthcare Institution "City Psychiatric Hospital No. 6 (Inpatient Department with Treatment Center), Saint Petersburg
  - 444-SPHI "City Mental Hospital #3 n.a. I.I.Skvortsov-Stepanov", Saint Petersburg
  - 452-Saint Petersburg State Public Institution of Healthcare "City Psychiatric Hospital #3 n.a. I. I. Skvortsov-Stepanov",, Saint Petersburg
  - 496-SPHI "City Mental Hospital #3 n.a. I.I.Skvortsov-Stepanov", Saint Petersburg
  - 458-State Budget Healthcare Institution "Samara Psychiatric Hospital, Samara
  - 416-FSBEI HE "Smolensk State Medical University" of the MoH of the RF (Clinical Research Centre of diagnostics and medicines), Smolensk
  - 572-Klinika StoLet" Ltd., Tomsk
  - 422-State Budget healthcare Institution of Yaroslavl region "Yaroslavl region clinical psychiatric hospital", Yaroslavl
- Serbia (10):
  - 424-Institute of Mental health, Belgrade
  - 425-Clinical Hospital Center "Dr. Dragisa Misovic-Dedinje", Clinic of Psychiatry, Belgrade
  - 584-Clinic for Psychiatry, Clinical Canter of Serbia, Belgrade
  - 587-Institute of Mental health, Belgrade
  - 472-Special Neuropsychiatric Hospital Kovin, Kovin
  - 430-Psychiatric Clinic, Clinical Center Kragujevac, Kragujevac
  - 423-Clinical Center Kragujevac, Clinic of Psychiatry, Kragujevac
  - 427-Clinical Center Nis, Mental Health Protection Clinic, Niš
  - 585-Special Hospital for Psychiatric Diseases "Gornja Toponica", Niš
  - 593-Specialized Hospital for Neuropsychiatric Diseases "Sveti Vracevi", Novi Kneževac
- Spain (8):
  - 574-Hospital Clinic de Barcelona, Barcelona
  - 576-Hospital Universitari Vall d'Hebron, Barcelona
  - 588-Institucion Hospitalaria Hestia Palau - Ensayos clinicos, Barcelona
  - 475-Hospital Gregorio Marañon, Madrid
  - 575-Hospital Universitario 12 de Octubre, Madrid
  - 494-CSM La Corredoria, Oviedo
  - 431-Hospital Psiquiátrico Provincial Doctor Villacian, Valladolid
  - 529-Hospital Provincial de Zamora, Zamora
- Ukraine (9):
  - 508-CI Cherkasy Regional Psychiatric Hospital of ChRC, Smila, Cherkasy Oblast
  - 564-Regional Clinical Psychiatric Hospital, Kropyvnytskyi, Kirovograd Region
  - 460-Kyiv City Psychoneurological Hospital #3 General Psychiatry Department No. 2, Kyiv, Vasylkiv District Kyiv Region
  - 434-State Institution "Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine", Department of Urgent Psychiatry and Narcology, Kharkiv
  - 567-"CIH Kharkiv Regional Clinical Psychiatric Hospital #3 Psychiatric Department of Primary Psychotic Episod Short Site name: CIH KRCPH #3 PD of PPE ", Kharkiv
  - 582-SI Institute of Neurology,Psychiatry&Narcology of NAMSU, Kharkiv
  - 435-Kyiv Regional Medical Incorporation "Psychiatry". Center of Novel Treatment and Rehabilitation of Psychotic disorders, build 5, Department #30, Kyiv
  - 565-"Kyiv CH on Railway Transport #2 of Branch Center of Healthcare Public Company Ukr Railway Short site name: Kyiv Railway Clinical Hospital № 2", Kyiv
  - 509-CI Odesa Regional Medical Centre of Mental Health, Odesa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Darwish M, Bugarski-Kirola D, Passarell J, Owen J, Jaworowicz D, DeKarske D, Stankovic S. Pimavanserin Exposure-Response Analyses in Patients With Schizophrenia: Results From the Phase 2 ADVANCE Study. J Clin Psychopharmacol. 2022 Nov-Dec 01;42(6):544-551. doi: 10.1097/JCP.0000000000001611. Epub 2022 Oct 3. PMID 36190440

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Drug - Pimavanserin | Placebo
Started | 227 | 226
Completed | 195 | 188
Not Completed | 32 | 38
Not completed — Withdrawal by Subject | 10 | 11
Not completed — Adverse Event | 6 | 14
Not completed — Protocol Violation | 6 | 9
Not completed — Non-compliance with study drug | 3 | 2
Not completed — Use of prohibited medication | 2 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Geopolitical conflict | 2 | 0
Not completed — Lack of Efficacy | 3 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug - Pimavanserin | Placebo | Total
Number analyzed (Participants) | 227 | 226 | 453
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 227 | 226 | 453
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 36.3 (9.61) | 37.5 (9.78) | 36.9 (9.71)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 90 | 185
  Male | 132 | 136 | 268
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 225 | 224 | 449
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Argentina | 39 | 39 | 78
  Hungary | 4 | 7 | 11
  Czechia | 3 | 7 | 10
  Ukraine | 23 | 21 | 44
  Poland | 6 | 2 | 8
  Italy | 2 | 3 | 5
  Bulgaria | 70 | 74 | 144
  Lithuania | 1 | 0 | 1
  Serbia | 21 | 24 | 45
  Croatia | 5 | 8 | 13
  Russia | 43 | 34 | 77
  Spain | 10 | 7 | 17
Negative Symptom Assessment-16 (NSA-16) [Mean (Standard Deviation); unit: Score] — The NSA-16 is a semi-structured interview and a validated scale containing 16 items for evaluating negative symptoms of schizophrenia, i.e. the reduction or absence of emotional expression and volitional behaviors normally present in a healthy person. Items are scored based on behaviors during the interview (items 1-4, 6, 7, 9, 11, 15, 16) or previous 7 days (items 5, 8, 10, 12-14) on a 6-point scale from 1 to 6. The NSA-16 total score is the sum of item scores. It can range from 16 to a maximum of 96, with higher scores denoting more severe negative symptoms in schizophrenia.
  Score | 61.3 (8.04) | 60.8 (7.86) | 61.1 (7.95)
CGI-SCH S of negative symptoms score [Mean (Standard Deviation); unit: Score] — The Clinical Global Impression of Schizophrenia Scale-Severity (CGI-SCH S) is a clinician-rated, 7-point scale to evaluate positive, negative, depressive, cognitive symptoms and overall severity in schizophrenia. For the purpose of this study, only the negative symptoms were evaluated. The score could range from 1 (normal, not ill) to 7 (among the most severely ill).
  Score | 4.8 (0.60) | 4.8 (0.57) | 4.8 (0.58)

OUTCOME MEASURES:

1. Primary Outcome: Negative Symptom Assessment-16 (NSA-16) Total Score - Change From Baseline to Week 26
Description: The NSA-16 is a semi-structured interview and a validated scale containing 16 items for evaluating negative symptoms of schizophrenia, i.e. the reduction or absence of emotional expression and volitional behaviors normally present in a healthy person. Items are scored based on behaviors during the interview (items 1-4, 6, 7, 9, 11, 15, 16) or previous 7 days (items 5, 8, 10, 12-14) on a 6-point scale from 1 to 6. The NSA-16 total score is the sum of item scores. It can range from 16 to a maximum of 96, with higher scores denoting more severe negative symptoms in schizophrenia.
Time Frame: 26 Weeks Treatment Duration
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug - Pimavanserin | Placebo
Number analyzed (Participants) | 224 | 222
score on a scale | -12.14 (10.29) | -11.09 (9.18)
Statistical Analysis 1: Comparison: Drug - Pimavanserin vs Placebo; Difference between LSM changes for adjunctive pimavanserin and adjunctive placebo (pimavanserin - placebo) at the specified visit from MMRM analysis; Test type: Superiority; p = 0.4825, Mixed Models Analysis — Two-sided p-value for treatment difference at Week 26 from MMRM analysis

2. Secondary Outcome: Clinical Global Impression of Schizophrenia Scale-Severity (CGI-SCH-S) of Negative Symptoms Score - Change From Baseline to Week 26
Description: The Clinical Global Impression of Schizophrenia Scale-Severity (CGI-SCH S) is a clinician-rated, 7-point scale to evaluate positive, negative, depressive, cognitive symptoms and overall severity in schizophrenia. For the purpose of this study, only the negative symptoms were evaluated. The score could range from 1 (normal, not ill) to 7 (among the most severely ill).
Time Frame: 26 Weeks Treatment Duration
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug - Pimavanserin | Placebo
Number analyzed (Participants) | 224 | 222
score on a scale | -0.88 (0.91) | -0.87 (0.92)
Statistical Analysis 1: Comparison: Drug - Pimavanserin vs Placebo; Test type: Superiority; p = 0.8872, Mixed Models Analysis — Two-sided p-value for treatment difference at Week 26 from MMRM analysis

ADVERSE EVENTS:
Time Frame: 26 weeks
Arm/Group | Drug - Pimavanserin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/227 | 0/226
Serious Adverse Events (participants affected / at risk) | 2/227 | 7/226
Other Adverse Events (participants affected / at risk) | 9/227 | 16/226
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug - Pimavanserin (N=227) | Placebo (N=226)
Schizophrenia (Psychiatric disorders) | 0 (0) | 4 (4)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0)
Irritability (Psychiatric disorders) | 0 (0) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Drug - Pimavanserin (N=227) | Placebo (N=226)
Headache (Nervous system disorders) | 9 (12) | 16 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-05): https://cdn.clinicaltrials.gov/large-docs/82/NCT04531982/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-11): https://cdn.clinicaltrials.gov/large-docs/82/NCT04531982/SAP_001.pdf